CLINICAL TRIAL: NCT02165488
Title: Gastrointestinal, Hepatic and Biliary Sequelae of Frequent Ketamine Use: a Prospective Observational Study
Brief Title: Frequent Ketamine Use and Gastrointestinal, Liver and Biliary Sequelae
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wai-Kay Seto, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: UW14-237
Record Dates: First submitted 2014-06-08; First posted 2014-06-17 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Gastritis; Peptic Ulcer Disease; Cholangiopathy; Liver Fibrosis
Keywords: ketamine; abuse; abdominal discomfort; cholangiopathy
MeSH Terms: conditions — Gastritis; Peptic Ulcer; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saved plasma samples Gastric antral and duodenal histology obtained by upper GI endoscopy
Oversight: Data Monitoring Committee: No

SUMMARY:
30% of ketamine users complain of abdominal discomfort. Long-term ketamine use is associated with hepatotoxicity and pathologic changes to the biliary tract. Yet the prevalence of gastrointestinal and hepatobiliary pathologies in ketamine users has not been well-described. The investigators plan to recruit a large number of ketamine users based on referrals from different Psychiatry clusters in Hong Kong and to investigate the underlying cause of abdominal discomfort, describe the prevalence of different gastrointestinal and hepatobiliary pathologies and describe their long-term outcome.

DETAILED DESCRIPTION:
The recreational use of psychotropic drugs has been increasing over the past 2 decades in Hong Kong. Ketamine hydrochloride is currently one of the most popular recreational drugs in Hong Kong, and its recreational use is also increasing in the United Kingdom and Europe. Inhalation of ketamine could result in hallucinations, out-of-the-body experiences and psychological dissociation, making it popular among young adults. One of the well-known side effects of ketamine is bladder dysfunction, which is seen in one-quarter of chronic ketamine users .

Ketamine has also been known to be associated with gastrointestinal symptoms. Colicky epigastric / abdominal discomfort in ketamine users, known as "K-cramps", has been reported in 33.3% of frequent ketamine users, and is the second-most common symptom of presentation (21%) among ketamine users in the emergency department . Nonetheless, the underlying etiology resulting in this abdominal discomfort remains poorly defined. A possible etiology is intestinal motility disorders, since ketamine interferes with gastric motility. Another possible cause could be ketamine-related cholangiopathy, which has been described in both Asia and Western countries. Another possible cause could be ketamine-related liver dysfunction, which is seen in 16% of ketamine users. Chronic ketamine hepatotoxicity is associated with mitochondrial liver injury , and could result in bridging liver fibrosis.

We plan to recruit subjects from ketamine users seeking medical attention at substance abuse clinics in different psychiatric clusters in Hong Kong. A screening log will be kept on the total number of ketamine users attending different substance abuse clinics and the number of potential subjects referred to our center.

Baseline sociodemographic information will be obtained. A standardized method will be used to assess and quantify the degree of ketamine use, as well as the recreational use of other psychotropic drugs (e.g. ecstasy, methamphetamine, marijuana etc.) and alcohol intake. Subjects will then be assessed for the presence or absence of dyspepsia, biliary-type abdominal pain， gastroparesis or other abdominal symptoms following standard criteria.

ELIGIBILITY:
Inclusion Criteria:

* Use of ketamine or ketamine mixed with other psychotropic drugs with frequency of at least twice per month over 6 months within the last 2 years.
* Recurrent abdominal discomfort over the past 3 months or more.
* Han Chinese ethnicity.
* Age 18-60 years.

Exclusion Criteria:

* Mental retardation or unable to give informed consent
* Co-existing biliary disorders including recurrent pyogenic cholangitis, primary sclerosing cholangitis, IgG4 sclerosing cholangiopathy and HIV cholangiopathy.
* Other significant medical co-morbidities

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Recreational use of ketamine with frequency at least twice per month over 6 months within the last 2 years, with or without other illicit psychotropic drug.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-06; Primary Completion 2019-05 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Incidence of cholangiopathic changes | 3 months
Incidence of peptic ulcer disease | 3 months
Incidence of liver fibrosis | 3 months

SECONDARY OUTCOMES:
Long-term outcome of peptic ulcer disease in ketamine users | 24 months
Long-term outcome of liver fibrosis in ketamine users | up to 24 months
Long-term outcomes of cholangiopathic changes in ketamine users | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Seto WK, Mak SK, Chiu K, Vardhanabhuti V, Wong HF, Leong HT, Lee PSF, Ho YC, Lee CK, Cheung KS, Yuen MF, Leung WK. Magnetic resonance cholangiogram patterns and clinical profiles of ketamine-related cholangiopathy in drug users. J Hepatol. 2018 Jul;69(1):121-128. doi: 10.1016/j.jhep.2018.03.006. Epub 2018 Mar 16. PMID 29551711